CLINICAL TRIAL: NCT00000975
Title: Pilot Study To Determine the Feasibility of Itraconazole for Primary Treatment and Suppression of Relapse of Disseminated Histoplasmosis in Patients With the Acquired Immunodeficiency Syndrome
Brief Title: A Study of Itraconazole in the Treatment and Prevention of Histoplasmosis, a Fungal Infection, in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 120; 11095 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Histoplasmosis
Keywords: AIDS-Related Opportunistic Infections; Histoplasmosis; Drug Evaluation; Antifungal Agents; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Histoplasmosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
To evaluate the feasibility of itraconazole as (1) primary therapy in histoplasmosis and (2) maintenance therapy after completion of primary therapy. To evaluate the effect of therapy of CNS histoplasmosis. To determine if resistance to drug occurs in patients who fail therapy.

Histoplasmosis is a serious opportunistic infection in patients with AIDS. Although the clinical response to amphotericin B treatment in the AIDS patients is generally good, administration difficulties and toxicity detract from its usefulness. Oral treatment with ketoconazole overcomes these limitations of amphotericin B, but does not appear to be effective for primary treatment in patients with AIDS. Itraconazole is a triazole compound in which preclinical studies have demonstrated activity against Histoplasmosis capsulatum. Preclinical studies have also shown that itraconazole appears effective in the treatment of histoplasmosis. The frequency of adverse reactions to itraconazole has been low in several studies. Central nervous system (CNS) involvement occurs in up to 20 percent of patients with histoplasmosis, and appears to have a poor response to amphotericin B treatment. Itraconazole has been used successfully in a small number of patients with cryptococcal meningitis, supporting a study of its use in CNS histoplasmosis.

DETAILED DESCRIPTION:
Histoplasmosis is a serious opportunistic infection in patients with AIDS. Although the clinical response to amphotericin B treatment in the AIDS patients is generally good, administration difficulties and toxicity detract from its usefulness. Oral treatment with ketoconazole overcomes these limitations of amphotericin B, but does not appear to be effective for primary treatment in patients with AIDS. Itraconazole is a triazole compound in which preclinical studies have demonstrated activity against Histoplasmosis capsulatum. Preclinical studies have also shown that itraconazole appears effective in the treatment of histoplasmosis. The frequency of adverse reactions to itraconazole has been low in several studies. Central nervous system (CNS) involvement occurs in up to 20 percent of patients with histoplasmosis, and appears to have a poor response to amphotericin B treatment. Itraconazole has been used successfully in a small number of patients with cryptococcal meningitis, supporting a study of its use in CNS histoplasmosis.

At least 30 patients with AIDS and an initial episode of disseminated histoplasmosis are selected for this study. Up to 5 patients will have a diagnosis of CNS histoplasmosis. Therapy with all other systemic antifungal agents must be halted before study entry. Patients receive itraconazole for 3 days followed by daily oral doses for a total of 12 weeks. Patients who are doing well clinically, without evidence of clinical failure or dose-limiting toxicity, are permitted to continue maintenance therapy to prevent relapse at a reduced dose for an additional 12 months. Patients who are being treated for CNS histoplasmosis will continue to receive itraconazole.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Vincristine, vinblastine, bleomycin, or interferon for Kaposi's sarcoma.
* Erythropoietin.
* Didanosine by exemption for 10 patients.
* Barbiturates.
* Coumarin-type anticoagulants.
* Oral contraceptives.
* Digoxin.
* Methadone.
* Narcotics.
* Acyclovir.
* Acetaminophen.
* Sulfonamides.
* Trimethoprim / sulfamethoxazole.
* Pentamidine for Pneumocystis carinii pneumonia (PCP) or PCP prophylaxis.
* Topical antifungals.
* Pyrimethamine.
* Ganciclovir.
* AZT.
* Stress doses of steroids in patients with adrenal insufficiency.

Concurrent Treatment:

Allowed:

* Dose reduction or interruption of myelosuppressive therapy and transfusion to maintain hemoglobin of 7 or more g/dl.
* Radiation therapy.

Patient must:

* Show laboratory evidence of HIV infection and disseminated histoplasmosis.
* Be oriented to person, place, and time.
* Be able to give written informed consent (appropriate consent must be obtained from a parent or legal guardian for patients under 18 years of age).

Allowed:

* Abnormal liver function tests in Grade 3 toxicity range if liver biopsy shows evidence that histoplasmosis caused these abnormalities.
* Mucocutaneous candidiasis.

Prior Medication:

Allowed:

* Amphotericin B or ketoconazole for pulmonary histoplasmosis at least 3 months prior to study entry.
* Azidothymidine (AZT).
* Vincristine, vinblastine, bleomycin, or interferon for mucocutaneous Kaposi's sarcoma.
* Prophylaxis for Pneumocystis carinii pneumonia (PCP).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Severely ill, or at risk of dying from histoplasmosis within the first week of treatment, as indicated by systolic blood pressure less than 90 mm Hg , or PO2 less than 60.
* Active CNS lesions, malignancies, or infections other than MAI.
* Severe malabsorption syndrome (persistent diarrhea more than 4 weeks duration with at least 4 loose stools per day accompanied by a 10 percent or greater weight loss).
* Requiring cytotoxic therapy for malignancies.
* Any systemic fungal infection other than histoplasmosis.
* Systemic Mycobacterium avium intracellulare.
* Receiving treatment for other acute opportunistic infections whose signs and symptoms have not yet resolved or stabilized.
* History of allergy to or intolerance of imidazoles or azoles.

Concurrent Medication:

Excluded:

* All other systemic antifungal agents.
* Investigational drugs not specifically allowed.
* Oral hypoglycemics.
* Rifamycins.
* Phenytoin.
* Carbamazepine.
* Steroids in excess of physiologic replacement doses not specifically allowed.
* Cytotoxic chemotherapy.
* Discouraged:
* Antacids.
* Sucralfate.
* H2 blockers.

Patients with the following are excluded:

* Severely ill, or at risk of dying from histoplasmosis within the first week of treatment.
* Active CNS infections, malignancies or lesions not documented to be caused by histoplasmosis, which would interfere with assessment of response.
* Unable to take oral medications reliably.
* Severe malabsorption syndrome.
* Requiring cytotoxic therapy for malignancies.
* Any systemic fungal infection other than histoplasmosis.
* Systemic Mycobacterium avium intracellulare.
* Receiving treatment for other acute opportunistic infections whose signs and symptoms have not yet resolved or stabilized.

Prior Medication:

Excluded for greater than 1 week within the last 3 months:

* Fluconazole.
* Itraconazole.
* SCH 39304.
* Amphotericin B greater than 1.5 mg/kg, or any other antifungal for this episode of disseminated histoplasmosis.

Patients who the investigator feels would be undependable with regard to adherence to the protocol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Study Completion 1994-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LJ Wheat, Study Chair
Locations (12):
- United States (12):
  - USC CRS, Los Angeles, California
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Hecht FM, Wheat J, Korzun AH, Hafner R, Skahan KJ, Larsen R, Limjoco MT, Simpson M, Schneider D, Keefer MC, Clark R, Lai KK, Jacobson JM, Squires K, Bartlett JA, Powderly W. Itraconazole maintenance treatment for histoplasmosis in AIDS: a prospective, multicenter trial. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Oct 1;16(2):100-7. doi: 10.1097/00042560-199710010-00005. PMID 9358104
- [Background] Wheat J, Hafner R, Korzun AH, Limjoco MT, Spencer P, Larsen RA, Hecht FM, Powderly W. Itraconazole treatment of disseminated histoplasmosis in patients with the acquired immunodeficiency syndrome. AIDS Clinical Trial Group. Am J Med. 1995 Apr;98(4):336-42. doi: 10.1016/s0002-9343(99)80311-8. PMID 7709945